CLINICAL TRIAL: NCT00731835
Title: Ischemic Foot Ulcers: Is Intervention Better Than Wound Care Alone? A Randomized Controlled Trial
Brief Title: Ischemic Foot Ulcers: Is Intervention Better Than Wound Care Alone
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment
Sponsor: University of Pittsburgh (Other)
Collaborators: Society for Vascular Surgery (Other)
Responsible Party: Principal Investigator, Rabih A. Chaer, Associate Professor of Surgery, University of Pittsburgh
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol #2, Version 1
Record Dates: First submitted 2008-08-06; First posted 2008-08-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Ischemic Foot Ulcer
Keywords: Vascular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (No Intervention): 1. Wound Care (group 1)--Best standard wound care with aggressive debridement
- Group 2 (Active Comparator): 2. Endovascular Intervention + Wound Care (group 2)--Best standard wound care in combination with endovascular revascularization
  Endovascular revascularization is the intervention
  Interventions: Procedure: Endovascular Revascularization

INTERVENTIONS:
Procedure: Endovascular Revascularization — * angioplasty, also called percutaneous transluminal angioplasty (PTA) and/or
  * stent placement
  * atherectomy
  Arms: Group 2

SUMMARY:
You are being asked to take part in this study because your doctor has determined that you have an ischemic foot ulcer. This research study will compare two approved standard of care treatment modalities for the management of ischemic foot ulcers. The ischemic foot ulcer (wound) on your foot is a result of a blocked artery in your leg. The wound can sometimes be healed with wound care alone, which includes dressing changes with creams and removing (debriding) the dead tissue. Alternatively, the significant narrowing or blockage in one of the arteries in your leg can be treated with several endovascular treatment techniques including:

* angioplasty, also called percutaneous transluminal angioplasty (PTA) and/or
* stent placement
* atherectomy

The hypothesis of this study is that early endovascular or surgical intervention in subjects with moderate arterial insufficiency and a non-healing foot ulcer results in a higher overall incidence of wound healing in a significantly shorter period of time.

DETAILED DESCRIPTION:
Design:

This study is a single center, prospective, randomized trial evaluating the benefit of endovascular intervention on the healing of ischemic foot ulcers when compared to best wound care alone. The study population will be comprised of subjects with a foot ulcer and non-palpable or diminished pedal pulses. The expected duration of subjects in this trial is 2 years.

Patients will be randomized into two groups:

1. Wound Care (group 1)--Best standard wound care with aggressive debridement
2. Endovascular Intervention + Wound Care (group 2)--Best standard wound care in combination with endovascular revascularization

Subjects will undergo standard of care evaluation for ischemic foot ulcers. These same evaluations would be performed whether or not the subject was participating in this research study. In the event that a clinically significant event or unanticipated disease or condition is identified, the subject and their doctor will be notified, the investigator, will review the results of the tests and procedures that are standard of care, and the results will become part of the research record. Prior to undergoing randomization, the subject will sign and fully understand an IRB consent form that is HIPAA compliant.

ELIGIBILITY:
Inclusion Criteria:

* The subject (male or non-pregnant female) must be greater than or equal to 18 years of age
* Ischemic ulcer of foot present
* An ankle-brachial index (ABI) of 0.4 to 0.8 or monophasic-biphasic waveforms on pulse volume recordings. (If the subject is diabetic or has renal failure, with incompressible vessels, a toe brachial index of 0.4 to 0.8 is required.)
* Signed informed consent

Exclusion Criteria:

* Severe ischemia as defined by advanced gangrene, an ABI of less then or equal to 0.3 and monophasic waveforms on pulse volume recording
* Advanced renal insufficiency, defined as serum creatinine greater than or equal to 3 mg/dl
* Absolute contraindication to contrast media, as determined by the investigator
* Unwilling or unable to provide informed consent or return for required follow-up evaluations.
* Previous enrollment in this clinical study
* Concurrent participation in another clinical research study

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Primary endpoint: wound healing at 4 weeks and 12 weeks | 4 weeks and 12 weeks

SECONDARY OUTCOMES:
Secondary endpoints: amputation free survival, time to healing, quality of life, major adverse events. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States